CLINICAL TRIAL: NCT02262052
Title: Advanced Diagnostic Management of Suspected Recurrent Ipsilateral Deep Vein Thrombosis of the Leg With Magnetic Resonance Direct Thrombus Imaging
Brief Title: Advanced Diagnostic Management of Suspected Recurrent Ipsilateral DVT With MRDTI
Acronym: Theia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Trombosestichting Nederland (Unknown)
Responsible Party: Principal Investigator, Erik Klok, Dr, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LeidenU
Record Dates: First submitted 2014-09-23; First posted 2014-10-10 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Diagnostic management; Recurrent; MRI; Ipsilateral
MeSH Terms: conditions — Venous Thrombosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 4 cohort study (Other): MRDTI
  Interventions: Other: MRDTI

INTERVENTIONS:
Other: MRDTI — MRDTI is primary diagnostic test for management of suspected ipsilateral DVT

SUMMARY:
The Theia-study is a prospective, multicenter, single-arm management (cohort) study.

Consecutive patients with clinically suspected acute, recurrent, ipsilateral, proximal deep vein thrombosis (DVT) of the leg, who fulfil all the inclusion criteria and meet none of the exclusion criteria, are eligible for inclusion and will be managed according to the result of a magnetic resonance direct thrombus imaging (MRDTI) of the affected leg. The MRDTI is to be performed and adjudicated within 24 hours of study inclusion. The final treatment decision will be made based on this ruling of the MRDTI. In case of a positive MRDTI signal, patients will be treated with therapeutically dosed anticoagulants or modified in patients with a recurrent DVT on anticoagulant therapy. Patients with a negative MRDTI ruling will be left untreated, or treatment will be remained unadjusted if they are on anticoagulant treatment at inclusion. All patients with negative MRDTI will be subjected to a standardized compression ultrasonography (CUS) within 48 hours after initial presentation. The latter CUS serves as a reference test in case the patient returns with symptoms of ipsilateral recurrence in the future, and will not be used for management decisions at baseline. The study flowchart can be found in Appendix A.

All patients will be followed for three months for the occurrence of acute recurrent venous thrombo-embolism (VTE). In case of suspected recurrent VTE, objective testing including either computed tomography pulmonary angiography (CTPA) for PE or CUS for DVT will be performed. Additionally, in case of a proven ipsilateral recurrent DVT during follow-up, MRDTI will be repeated.

DETAILED DESCRIPTION:
See below.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand the character and individual consequences of this study;
2. Signed and dated informed consent of the subject available before the start of any specific study procedures;
3. Age ≥18 years;
4. Suspected acute recurrent ipsilateral DVT, as defined by a documented prior objectivated episode of DVT in the same leg as current symptoms originate from

Exclusion Criteria:

1. General contraindications for MRI: claustrophobia, pregnancy, intracranial vascular clips, any ferromagnetic implants, presence of a cardiac pacemaker or defibrillator, metallic splinters in the eye, any trauma or surgery which may have left ferromagnetic material in the body;
2. CUS-proven acute symptomatic DVT within 6 months before current presentation;
3. Onset of symptoms suggestive of acute recurrent DVT more than 10 days prior to presentation;
4. Suspected acute PE;
5. Hemodynamic instability at presentation (as a consequence of concurrent acute PE or otherwise);
6. Medical or psychological condition that would not permit completion of the study or signing of informed consent, including life expectancy less than 3 months, or unwillingness to sign informed consent;
7. Non-compliance or inability to adhere to treatment or follow-up visits.
8. Patients with suspected acute, recurrent, ipsilateral DVT on therapeutic anticoagulant treatment > 48 hours at inclusion*

Note: *From August 2015 onward, patients with suspected acute, recurrent, ipsilateral DVT on anticoagulant treatment were allowed in the study as they were found to represent a high proportion (30%) of the screened study population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
3-month incidence of recurrent VTE in patients with negative MRDTI | 3-month follow-up
  Primary outcome is subdivided in two main outcomes: 3-month incidence of recurrent VTE in 1) patients with negative MRDTI for both DVT and thrombophlebitis who were not treated with any anticoagulant during follow-up and 2) all patients with negative MRDTI for DVT; these recurrences need to be objectively confirmed by either CT (for acute PE), or CUS with the baseline CUS serving as reference.

SECONDARY OUTCOMES:
3-month incidence of recurrent VTE in patients with normal D-dimer test and unlikely clinical probability according to the Wells clinical decision rule for DVT | 3-month follow-up
  the 3-month incidence of recurrent VTE in patients with low probability Wells score and a normal D-dimer test at baseline

OTHER OUTCOMES:
The feasibility of MRDTI in day to day clinical practice | First 24 hours after presentation to the emergency ward (post-hoc analysis)
  The feasibility of MRDTI in day to day clinical practice: percentage of eligible patients that had to be excluded due to logistic reasons such as unavailability of MRDTI within 24 hours of presentation.
Inter-observer variability of MRDTI | After the study has been completed, all MRDTI studies will be re-evaluated (post-hoc analysis)
  The inter-observer variability of MRDTI in daily clinical practice: all MRDTI scans will be review post-hoc by two independent experts to determine the alpha statistic between the readings in clinical practice and that by experts.
a formal cost-effectiveness and cost-utility analysis | This model will be based on the primary and secondary endpoints, scored after a follow-up period of 3 months (post-hoc analysis)
  A Markov model will be developed to estimate the cost-effectiveness MRDTI versus ultrasonography. The model will follow the patients through the course of disease in a maximum of two three-month cycles, and will include all relevant clinical outcomes and incorporated health states stratified by diagnostic management. Clinical events included in the model are fatal PE, recurrent VTE, major bleeds and clinically relevant non-major. The model includes clinical and cost outcomes, along with incremental cost-effectiveness ratios (ICERs) and net monetary benefits (NMBs).

CONTACTS AND LOCATIONS:
Overall Officials: F.A. Klok Klok, MD PhD, Principal Investigator — Department of Thrombosis and Hemostasis, LUMC, Leiden; M.V. Huisman, Prof, Principal Investigator — Department of Thrombosis and Hemostasis, LUMC, Leiden; L.J.M. Kroft, MD PhD, Principal Investigator — Department of Radiology, LUMC, Leiden
Locations (12):
- Ottawa Hospital, Ottawa, Canada
- RAMBAM Healthcare center, Haifa, Israel
- Netherlands (8):
  - AMC, Amsterdam
  - Rijnstate, Arnhem
  - Deventer Ziekenhuis, Deventer
  - LUMC, Leiden
  - HAGA, The Hague
  - MCH Westeinde, The Hague
  - Diakonessenhuis Utrecht, Utrecht
  - UMCU, Utrecht
- Ostfold Hospital Trust, Grålum, Norway
- Danderyds sjukhus, Stockholm, Sweden

REFERENCES:
- [Result] Tan M, Mol GC, van Rooden CJ, Klok FA, Westerbeek RE, Iglesias Del Sol A, van de Ree MA, de Roos A, Huisman MV. Magnetic resonance direct thrombus imaging differentiates acute recurrent ipsilateral deep vein thrombosis from residual thrombosis. Blood. 2014 Jul 24;124(4):623-7. doi: 10.1182/blood-2014-04-566380. Epub 2014 Jun 13. PMID 24928859
- [Result] Westerbeek RE, Van Rooden CJ, Tan M, Van Gils AP, Kok S, De Bats MJ, De Roos A, Huisman MV. Magnetic resonance direct thrombus imaging of the evolution of acute deep vein thrombosis of the leg. J Thromb Haemost. 2008 Jul;6(7):1087-92. doi: 10.1111/j.1538-7836.2008.02986.x. Epub 2008 Jul 1. PMID 18433464
- [Derived] van Dam LF, Dronkers CEA, Gautam G, Eckerbom A, Ghanima W, Gleditsch J, von Heijne A, Hofstee HMA, Hovens MMC, Huisman MV, Kolman S, Mairuhu ATA, Nijkeuter M, van de Ree MA, van Rooden CJ, Westerbeek RE, Westerink J, Westerlund E, Kroft LJM, Klok FA; Theia Study Group. Magnetic resonance imaging for diagnosis of recurrent ipsilateral deep vein thrombosis. Blood. 2020 Apr 16;135(16):1377-1385. doi: 10.1182/blood.2019004114. PMID 32016390